CLINICAL TRIAL: NCT06162663
Title: Double-blind Randomized Controlled Trial Comparing Suvorexant 20 mg to Placebo for Treatment of Insomnia in Cancer Survivors
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Sarah Tucker Marrison, Assistant Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Pro00130637
Record Dates: First submitted 2023-11-29; First posted 2023-12-08 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Insomnia
MeSH Terms: conditions — Breast Neoplasms; Sleep Initiation and Maintenance Disorders | interventions — suvorexant

STUDY DESIGN:
Intervention Model Description: Randomized double blind placebo controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Suvorexant with information on sleep hygiene (Experimental): Participants randomized to this arm will receive 10 mg of suvorexant daily with a dose increase to 20 mg after day 7. Medication will be administered as an oral medication. Total duration of 28 days.
  Interventions: Drug: Suvorexant Tablets
- Placebo with information on sleep hygiene (Placebo Comparator): Participants randomized to this arm will receive 10 mg of suvorexant daily with a dose increase to 20 mg after day 7. Medication will be administered as an oral medication. Total duration of 28 days.
  Interventions: Other: Placebo Control

INTERVENTIONS:
Drug: Suvorexant Tablets — Suvorexant initially with 10-20 mg for 28 days
  Arms: Suvorexant with information on sleep hygiene
Other: Placebo Control — Matched Placebo Control for 28 days
  Arms: Placebo with information on sleep hygiene

SUMMARY:
Investigators propose a double-blind, placebo-controlled trial evaluating the use of the use of Suvorexant in breast cancer survivors on selective estrogen receptor modulators or aromatase inhibitors with sleep disturbance to assess the impact on insomnia symptoms and quality of life. Breast cancer survivors have an increased risk of insomnia for which Suvorexant has the has the potential ability to impact to improve sleep related outcomes and cancer survivorship outcomes. Breast cancer survivors with sleep disturbance based on an Insomnia Severity Index Score (ISI) >15 will be randomized to either Suvorexant or placebo, with both arms receiving education on sleep hygiene.

DETAILED DESCRIPTION:
Cancer survivors have an incidence of sleep disturbance and insomnia higher than the general population, with significant potential implications on health outcomes including in survivorship domains and mortality outcomes. Available pharmacologic options for management of sleep disturbance are limited in efficacy and in their side effects. Investigators propose a double-blind placebo-controlled trial evaluating the use of the use of Suvorexant in breast cancer survivors on selective estrogen receptor modulators or aromatase inhibitors with sleep disturbance to assess the impact on insomnia symptoms and quality of life. Evaluation of breast cancer survivors on endocrine therapy uses a study population with high 5-year survival rate while retaining the capacity for recruitment and creating an opportunity to explore potential effects on vasomotor symptoms. Suvorexant has the potential to have a significant impact in cancer survivors not only on sleep related outcomes but also on cancer survivorship outcomes.

The purpose of the research study is to evaluate the ability of Suvorexant, a medication approved by the Food and Drug Administration (FDA) for insomnia, to treat sleep disturbance in breast cancer survivors on endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult post menopausal breast cancer survivors (female, > 18 years old)
* current selective estrogen modulator or aromatase inhibitor use
* at least 6 weeks beyond completion of definitive treatment for breast cancer
* less than 5 years from time of diagnosis.

Exclusion Criteria:

* less than 6-month life expectancy
* current steroid use
* severe depression or anxiety
* severe hepatic impairment
* concurrent use of moderate or strong CYP3A inhibitors
* current receipt of hospice care
* severe mental illness
* current use of greater than 40 morphine milligram equivalents daily
* diagnosis of obstructive sleep apnea, narcolepsy or other sleep related illness other than insomnia
* pregnancy
* treatment with alternate pharmacotherapy for insomnia at the time of trial initiation
* menstrual cycle within the past year

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult women with history of breast cancer on a selective estrogen modulators or aromatase inhibitors with symptoms of insomnia as characterized by an ISI score of 15 or more will be included in the study population.
Enrollment: 44 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Participant reported insomnia symptoms evaluated using the Insomnia Severity Index (ISI) | Assessed at baseline, 2 weeks, 4 weeks
  The within-person change in Insomnia Severity Index (ISI) will be evaluated from baseline to 4 weeks. The ISI is a scored on a scale of 0-28 based on responses to 7 questions. Higher values indicate more severe symptoms of sleep disturbance.

SECONDARY OUTCOMES:
Vasomotor Symptoms assessed using the Hot Flash Related Daily Interference Scale | Assessed at baseline, 2 weeks, 4 weeks
  Evaluation of Vasomotor Symptoms by the hot flash related daily interference scale. The hot flash related daily interference scale ranges from 0-100 with higher scores indicated a greater level of interference.
Quality of Life evaluated using the SF-36 | Assessed at baseline, 4 weeks
  Evaluation using the SF-36. The SF-36 evaluates 8 multi-item scales (Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, Mental Health). Scores for each of these scales is 0-100 with higher scores indicated a higher health care related quality of life.
Quality of Life evaluated using the Cancer Problems in Living Scale (CPIL) | Assessed at baseline, 4 weeks
  Evaluation using the Cancer Problems of Living (CPIL) Scale. The CPIL includes multi-item list of problems for which the participant classifies each problem based on severity.
Pain Evaluation evaluated using the Brief Pain Inventory (BPI) | Assessed at baseline, 2 weeks, 4 weeks
  Evaluation conducted using the Brief Pain Inventory (BPI). Participants are asked to rate their current symptoms, their average experiences of pain, and the minimum and maximum intensities of their symptoms on scales that range from 0 to 10. A total pain severity score can be found by averaging these items. Higher scores indicated increased symptoms.
Medication Adherence | Assessed at baseline, 4 weeks
  Evaluated using the simplified medication adherence questionnaire (SMAQ). The Simplified Medication Adherence Questionnaire (SMAQ) is a short questionnaire posed directly to the participant regarding medication-taking habits composed of 6 multiple choice questions. Positive responses or more than 2 reported missed doses over the past week indicates medication non-adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Marrison, MD PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- MUSC Department of Family Medicine, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No